CLINICAL TRIAL: NCT06812936
Title: A Randomized Clinical Trial of the Effectiveness of Acupressure in Relieving Orthodontic Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ayat M. Hussein, Principal Investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 911424
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Orthodontic Pain (D013850); Pain Management (D016146); Acupressure (D056351); Analgesics, Non-Narcotic (D000700); Acetaminophen (D000082)
Keywords: Orthodontic Pain; Pain Management; Acupressure Therapy; Acetaminophen (Paracetamol); Nonpharmacological Pain Relief; Orthodontic Treatment; Fixed Orthodontic Appliances; Visual Analog Scale (VAS)
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Acupressure

STUDY DESIGN:
Intervention Model Description: This randomized, parallel-group, single-center clinical trial compares the effectiveness of acupressure versus acetaminophen in managing orthodontic pain after initial archwire placement. Patients will be randomly assigned (1:1) to either the acupressure or acetaminophen group. Pain perception will be assessed using the Visual Analog Scale (VAS) over five days. The study employs single blinding, where investigators assessing outcomes are masked to group allocation. Randomization is conducted using a computer-generated sequence. This study aims to determine whether acupressure can be a viable alternative to analgesic medication for orthodontic pain management.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study, investigators and outcomes assessors will be blinded to the intervention groups to minimize bias. The investigators responsible for data collection and pain assessment will not know whether participants received acupressure or acetaminophen. Similarly, the outcomes assessors analyzing the Visual Analog Scale (VAS) scores will be blinded to the group assignments to ensure unbiased statistical analysis. However, due to the nature of the interventions, participants cannot be blinded, as they will actively perform acupressure or take acetaminophen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen Group (Active Comparator): Participants in this group will be instructed to take acetaminophen 500mg, up to three times within the first 24 hours following the insertion of the archwire. The purpose of this intervention is to alleviate pain associated with orthodontic treatment. The analgesic effect of acetaminophen, which acts centrally to reduce pain, will be evaluated based on self-reported pain levels recorded using a visual analog scale (VAS) over the five-day post-bonding period.
  Interventions: Drug: Acetaminophen
- Acupressure Group (Experimental): Participants in this group will be instructed on how to apply acupressure to two specific points: the Jaw Chariot (St 6) and Facial Beauty (St 36). They will be guided to apply firm pressure to these points up to five times within the first 24 hours after archwire insertion to alleviate pain associated with orthodontic treatment. The effectiveness of acupressure in pain management will be evaluated based on self-reported pain levels recorded using a visual analog scale (VAS) over the first five days post-bonding. If pain persists, participants may use acetaminophen as a supplementary pain management option.
  Interventions: Procedure: Acupressure

INTERVENTIONS:
Drug: Acetaminophen — This intervention involves the administration of acetaminophen 500mg tablets, taken up to three times within the first 24 hours following archwire insertion to manage pain associated with orthodontic treatment. Acetaminophen is a centrally acting analgesic that reduces pain without significantly affecting tooth movement, making it a preferred choice for pain relief in orthodontic patients. Participants will be instructed to record their pain levels using a visual analog scale (VAS) over a five-day period post-bonding to assess the effectiveness of this treatment."
  Other Names: Paracetamol 500mg
  Arms: Acetaminophen Group
Procedure: Acupressure — This intervention involves the application of acupressure to two specific acupressure points: Jaw Chariot (St 6) and Facial Beauty (St 36). Participants will be trained to apply firm pressure to these points up to five times within the first 24 hours after archwire insertion to alleviate orthodontic pain. Acupressure is a non-invasive therapy based on traditional Chinese medicine that aims to stimulate the body's natural healing processes and promote pain relief by balancing energy flow. Participants will be instructed to record their pain levels using a visual analog scale (VAS) over the first five days post-bonding to assess its effectiveness.
  Arms: Acupressure Group

SUMMARY:
Orthodontic treatment with fixed appliances often causes pain, which peaks within 24 hours after archwire placement and lasts for several days. Patients commonly use analgesics such as acetaminophen to relieve pain, as it has minimal impact on tooth movement compared to NSAIDs. However, nonpharmacological approaches, such as acupressure, may offer an alternative method for pain relief. Acupressure is a traditional Chinese medicine technique that involves applying pressure to specific points on the body to reduce pain and promote relaxation.

This randomized clinical trial aims to compare the effectiveness of acupressure versus acetaminophen in relieving orthodontic pain during the first five days after initial archwire placement.

Study Design and Methodology

* A parallel-group, single-center, blinded, randomized trial at Almina Dental Clinics.
* Participants will be randomly assigned to one of two groups (1:1 ratio):

  1. Acetaminophen Group: Participants will take 500 mg of acetaminophen up to three times in the first 24 hours after archwire insertion.
  2. Acupressure Group: Participants will apply pressure on two acupressure points (St 6 and St 3) up to five times in the first 24 hours. If pain persists, they may take acetaminophen.
* Pain levels will be recorded using a Visual Analog Scale (VAS) twice daily for five days.
* The Mann-Whitney U test will be used to compare pain scores between groups.

Eligibility Criteria

Inclusion Criteria:

* Patients aged 12 years and older with full permanent dentition (excluding third molars).
* Undergoing fixed orthodontic treatment for the first time.
* Minimum crowding of 4 mm according to Little's Irregularity Index.
* No systemic diseases, periodontal diseases, or acute/chronic oral pain.

Exclusion Criteria:

* Chronic use of analgesic medications.
* Allergy or contraindications to acetaminophen.
* Pregnant patients or those with cleft lip/palate.
* Recent toothache or requiring tooth extractions.
* Female patients during their menstrual period.

Study Significance

This study evaluates whether acupressure can be an effective, nonpharmacological alternative to acetaminophen for managing orthodontic pain. If proven effective, acupressure could offer a safe, noninvasive method for pain relief with fewer side effects.

Ethical Considerations & Dissemination

* The study protocol will be reviewed and approved by an ethics committee.
* The research is self-funded.
* Results will be published in a scientific journal to contribute to orthodontic pain management research.

DETAILED DESCRIPTION:
Introduction

Orthodontic treatment with fixed appliances is often associated with pain and discomfort, peaking within the first 24 hours after archwire placement and gradually subsiding over five to six days. This pain is caused by pressure-induced ischemic changes in the periodontal ligament, leading to sterile necrosis and inflammation. The release of biochemical mediators such as prostaglandins, histamine, serotonin, and bradykinin contributes to the sensation of pain.

Pharmacological interventions, such as nonsteroidal anti-inflammatory drugs (NSAIDs) and acetaminophen, are the most commonly used pain management methods. However, NSAIDs can slow tooth movement by inhibiting prostaglandin synthesis, while acetaminophen, though considered safer, may still cause adverse reactions in some individuals. Given these concerns, nonpharmacological pain relief methods, such as acupressure, have gained interest.

Acupressure is a mechanical technique rooted in traditional Chinese medicine, where pressure is applied to specific acupoints to promote circulation, reduce muscle tension, and stimulate the body's natural pain-relieving mechanisms. Unlike acupuncture, which involves the insertion of needles, acupressure is a noninvasive therapy that can be easily self-administered. Studies have explored its effectiveness in various medical and dental conditions, but its role in orthodontic pain management remains under-researched.

Study Objectives

The primary objective of this study is to compare the effectiveness of acupressure versus acetaminophen in reducing pain following initial archwire placement. The study will measure pain perception using a visual analog scale (VAS) over the first five days of orthodontic treatment.

Study Design and Methodology

This study is a randomized, parallel-group, single-center clinical trial with an equal allocation ratio (1:1). The trial will be conducted in a private orthodontic clinic, involving 60 patients aged 12 years and older who are undergoing fixed orthodontic treatment.

Eligibility Criteria

Inclusion Criteria:

* Patients undergoing comprehensive fixed orthodontic treatment for the first time.
* Presence of a minimum of 4 mm crowding, with no impactions or unerupted teeth.
* No history of systemic or periodontal diseases.
* No acute or chronic pain in the oral cavity at the time of enrollment.
* No history of cleft lip, cleft palate, or recent tooth extractions.
* Female patients must not be in their menstrual period at the time of the study.

Exclusion Criteria:

* Patients using analgesic medications chronically or requiring prophylactic antibiotics.
* Patients currently taking analgesics or antibiotics.
* Patients with contraindications to acetaminophen, such as hypersensitivity or liver disease.
* Patients with a recent history of toothache.
* Pregnant patients.

Randomization and Blinding

Participants will be randomly assigned to one of two intervention groups using a computer-generated randomization sequence. Blinding will be applied to data collection and analysis, although blinding of the operator during acupressure instruction may not be feasible.

Intervention Groups

* Acetaminophen Group: Patients will take 500 mg of acetaminophen up to three times within the first 24 hours after archwire placement to manage pain.
* Acupressure Group: Patients will be instructed on how to apply acupressure to two key points for pain relief:

  1. Jaw Chariot (St 6): Located on the jaw muscle in front of the earlobe.
  2. Facial Beauty (St 3): Positioned at the bottom of the cheekbone below the pupil.

Patients will be guided to press these acupoints firmly while taking deep breaths for one minute, repeating the process up to five times within 24 hours. If pain persists, acetaminophen will be allowed as a rescue medication.

Outcome Measurement Pain levels will be assessed using a 10-point VAS, with scores recorded twice daily for five days following archwire placement, except on the first day, where pain is recorded once.

Sample Size Calculation

The sample size was determined based on previous studies, with a mean difference in VAS scores of 2 units (20%) and a standard deviation of 2.42. A total of 48 patients (24 per group) was required to achieve 80% power with a 0.05 alpha level. To account for dropout, the sample size was increased to 56 patients.

Stopping Rules

If a participant experiences severe pain beyond their tolerance threshold, the study will be terminated for that individual.

Data Management and Analysis

Data will be analyzed using SPSS version 25.0 for Windows.

Descriptive Statistics:

* Frequencies, percentages, means, medians, interquartile ranges, and standard deviations.

Inferential Statistics:

* The Mann-Whitney U test will compare pain scores between groups.

Ethical Considerations

The study protocol will be submitted for approval by an ethics committee. Informed consent will be obtained from all participants, and parental consent will be required for patients under 18.

Budget and Funding

This study is self-funded.

Conclusion

This study aims to provide valuable insights into the effectiveness of acupressure as a nonpharmacological pain management strategy in orthodontic treatment. If acupressure proves to be an effective alternative to acetaminophen, it could offer a safer, non-invasive option for managing orthodontic pain, reducing reliance on analgesic medications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have agreed to the research procedures and signed an informed consent form.
2. Upper and lower comprehensive fixed orthodontic appliances (with no history of previous orthodontic treatment).
3. They have a minimum crowding of 4mm according to Little's irregularity index (with no impactions/unerupted teeth).
4. Patients with no systematic/periodontal diseases.
5. If tooth extraction is needed, it is performed at least two weeks before fixed appliance placement or delayed after the study is completed.
6. Patients aged 12 years and above with full permanent dentition (excluding the third molars)
7. No current acute or chronic pain in the oral cavity.

Exclusion Criteria:

1. Patients who have been using analgesic medications chronically or require prophylactic antibiotic coverage.
2. Patients who are currently taking analgesics or antibiotics.
3. Female patients being in the menstrual period.
4. Patients with contraindications to the use of paracetamol (Hypersensitivity or anaphylaxis to any acetaminophen-like or -containing agents, in conjunction with alcohol, and patients with severe liver disease).
5. Patients who have recently experienced a toothache.
6. Patients who have a cleft lip or palate.
7. Pregnant patients.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparative Evaluation of Acetaminophen and Acupressure for Pain Management in Orthodontic Treatment | From archwire insertion to 5 days post-bonding
  This study aims to compare the effectiveness of two pain management methods-acetaminophen (500mg) and acupressure-following the insertion of an archwire in orthodontic patients. Pain perception will be measured using a Visual Analog Scale (VAS), where patients rate their pain on a scale from 0 (no pain) to 10 (worst possible pain). The study will assess pain relief over the first five days post-treatment, with pain levels recorded twice daily on days 2 to 5, and once on day 1. Patients will either take acetaminophen or perform acupressure on specific points of the body (St 6 and St 36) to relieve discomfort. The goal is to determine which method provides more effective pain relief during the early stages of orthodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yassir Abdulkadhim Professor Dr. Yassir Abdulkadhim Yassir, Ph.D. (Orthodontics) (UK), Study Director — University of Baghdad; Rawof R. Al Tuma, Ph.D. (Orthodontics), Study Director — College of Dentistry, University of Karbala, Iraq
Locations (1):
- Almina Dental Clinics., Karbala, Karbala Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YW, Wang HH. The effectiveness of acupressure on relieving pain: a systematic review. Pain Manag Nurs. 2014 Jun;15(2):539-50. doi: 10.1016/j.pmn.2012.12.005. Epub 2013 Feb 15. PMID 23415783
- [Background] • Gach, M.R. (1990). Acupressure's potent points: A guide to self-care for common ailments, 1st ed., Bantam.